CLINICAL TRIAL: NCT01407627
Title: Evaluation of Fructose Ingestion and the Renin Angiotensin System in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Sofia Ahmed, Dr. Sofia Ahmed, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: UCalgary Sugar Study; AIHS (Other Grant/Funding Number: Establishment Grant); University of Calgary (Other Grant/Funding Number: Dept of Med Developmental Fund)
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease
Keywords: human; fructose; dextrose; renin angiotensin system; kidney; renal hemodynamics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Fructose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fructose First (Experimental): 1. Study Day 1 - measurement of renal hemodynamics and blood pressure
  2. Subjects will ingest fructose 200g daily x 14d
  3. Study Day 2 - measurement of renal hemodynamics
  4. Minimum 1 week "washout" period
  5. Subjects will ingest dextrose 200g daily x 14d
  6. Study Day 3 - measurement of renal hemodynamics and blood pressure
  Interventions: Dietary Supplement: Fructose
- Dextrose First (Active Comparator): 1. Study Day 1 - measurement of renal hemodynamics and blood pressure
  2. Subjects will ingest dextrose 200g daily x 14d
  3. Study Day 2 - measurement of renal hemodynamics
  4. Minimum 1 week "washout" period
  5. Subjects will ingest fructose 200g daily x 14d
  6. Study Day 3 - measurement of renal hemodynamics and blood pressure
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Fructose — Subjects will be randomized to one of 2 sequences:
  Sequence 1: Fructose (intervention) 200g daily x 14d followed by Dextrose (control) 200g daily x 14d Sequence 2: Dextrose (control) 200g daily x 14d followed by Fructose (intervention) 200g daily x 14d

SUMMARY:
Fructose is an ingredient that is added to many of our foods. It is a cheaper, sweeter additive that can be found in everything from soda pop to yogurt to granola bars. In the last few years a significant number of studies have been published linking consumption of fructose with obesity, hypertension and more recently, kidney and cardiovascular disease.

Animal studies show a strong link between excessive ingestion of fructose and the development of kidney and cardiovascular disease mediated by the renin angiotensin system, a hormonal system whose activation is detrimental to both the kidney and the heart. There has been very little research done on the potentially pathophysiological relationship between a high fructose diet and kidney and cardiovascular disease in humans.

The investigators hypothesize that ingestion of fructose will result in upregulation of the renin angiotensin system in humans.

Cardiovascular disease in women is a significant risk factor. By having women participate who are on the birth control pill and as well as women who use non oral forms of birth control or no birth control, kidney function and cardiovascular health can be examined as it relates to in the influence oral hormones might play. How the kidney responds to the influence of sugar and fructose while a woman is on an oral birth control pill, may reveal mechanisms that could help us understand cardiovascular disease in women.

DETAILED DESCRIPTION:
PRIMARY AIM: To examine whether the physiologic and molecular responses to Angiotensin II (AngII) challenge differ in response to fructose intake as assessed by two independent means:

1. The renal and mean arterial pressure (MAP) response to an AngII challenge.
2. Reactive changes in circulating levels of renin and aldosterone with graded AngII challenge.

PRIMARY HYPOTHESES: Ingestion of fructose in healthy subjects will result in:

1. A decrease in renal and systemic sensitivity to infused AngII.
2. A decrease in the reactive changes in renin and aldosterone with graded AngII challenge.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years,
* able to comprehend study and comply with high-salt diet
* kidney disease (on the approval of their nephrologist)
* on an oral birth control pill and non oral birth control and those not on birth control

Exclusion Criteria:

* cardiovascular disease (symptoms consistent with myocardial ischemia, previously documented myocardial ischemia, cardiac arrhythmias or valve abnormalities, or abnormal ECG at screening)
* cerebrovascular disease (transient ischemic attacks or stroke)
* hypertension (BP>140/90 or use of antihypertensive medications)
* diabetes mellitus (defined by history, use of hypoglycemic agents or a fasting glucose >7mmol/L)
* hyperlipidemia (LDL >4.5mmol/L or use of lipid-lowering agents)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in filtration fraction | after 2 weeks of ingestion of fructose compared to baseline value
  To examine whether the physiologic and molecular responses to an Angiotensin II challenge differ in response to fructose intake as assessed by reactive changes in circulating levels of renin and aldosterone with a graded Angiotensin II challenge.

SECONDARY OUTCOMES:
change in blood pressure in response to angiotensin II challenge | change after 2 weeks of fructose ingestion
  To examine whether the physiologic and molecular responses to an Angiotensin II challenge differ in response to fructose intake as assessed by renal and mean arterial pressure (MAP) response to an Angiotensin II challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia B Ahmed, MD MMSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No